CLINICAL TRIAL: NCT02238522
Title: Phase 1 Open-label Dose Escalation and Expansion Study of ZEN003365 in Subjects With Relapsed or Refractory Lymphoproliferative Malignancies or Acute Myeloid Leukemia
Brief Title: Phase 1 Study Evaluating ZEN003365 in Relapsed/Refractory Lymphoproliferative Malignancies or Relapsed/Refractory AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Zenith Epigenetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEN-ONC3365-101
Record Dates: First submitted 2014-08-28; First posted 2014-09-12 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Lymphoproliferative Malignancies; Acute Myeloid Leukemia
Keywords: Chronic lymphocytic leukemia; B-prolymphocytic leukemia; Non-Hodgkin's lymphoma; follicular lymphoma; mantle cell lymphoma; marginal zone lymphoma; small lymphocytic lymphoma; diffuse large B-cell lymphoma; unclassifiable lymphoma; T-cell lymphoma; Richter's syndrome; Waldenström's macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation Stage - ZEN003365 (Experimental): ZEN003365 will be administered orally as a single agent, enrolling LPM patients and AML patients
  Interventions: Drug: ZEN003365
- Dose Expansion Stage - ZEN003365 (Experimental): ZEN003365 will be administered orally as a single agent, enrolling LPM patients and AML patients
  Interventions: Drug: ZEN003365

INTERVENTIONS:
Drug: ZEN003365

SUMMARY:
The purpose of this study is to determine safety, tolerability, dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of ZEN003365 in patients with relapsed/refractory lymphoproliferative malignancies (LPM) or relapsed/refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation and Expansion Stages:

* ECOG performance status ≤ 1 for LPM patients, ≤ 2 for AML patients
* Age 18 years or older
* Adverse events (AEs), except for alopecia, from any previous treatments must have recovered to eligibility levels from prior toxicity
* Adequate renal, hepatic and coagulation function, as specified per protocol
* Written informed consent granted prior to any study-specific screening procedures

LPM Patients:

* Histologically confirmed lymphoproliferative malignancy
* Have received prior protocol-specified disease-dependent prior treatments
* Have measurable disease
* Platelets ≥ 75,000/µL (≥50,000/µL if bone marrow involvement), absolute neutrophil count (ANC) ≥ 1,000/ µL, and hemoglobin (Hgb) ≥ 8 g/dL
* Patients must have been off previous anticancer therapy for at least 3 weeks or 5 half-lives, whichever is longer, and the subject must have recovered to eligibility levels from prior toxicity

AML:

* Refractory or relapsed AML patients, without curative intent, e.g., not a stem cell transplant candidate
* Any prior chemotherapy must have been completed ≥ 2 weeks, any therapy with biologics must have been completed ≥ 4 weeks prior to day 1 of study treatment, and the participant must have recovered to eligibility levels from prior toxicity
* Blast count ≤ 10,000/µL prior to initiation of therapy

Exclusion Criteria

Dose Escalation and Expansion Stages:

* Prior exposure to a BET inhibitor
* Prior allogeneic hematopoietic cell transplant
* Chronic graft versus host disease
* Known, active fungal, bacterial, and/or viral infection
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Current subdural hematoma
* CNS or leptomeningeal metastases
* Requirement for medications or agents known to be sensitive CYP3A4 substrate drugs, CYP3A4 substrate drugs with a narrow therapeutic range or to be strong inhibitors/inducers of CYP3A4
* Requirement for immunosuppressive agents
* Evidence of significant cardiovascular disease or significant screening ECG abnormalities
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient.

AML patients:

* Acute promyelocytic leukemia (APL)
* Chronic myeloid leukemia (CML) in blast crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Dose escalation stage - The safety of orally administered ZEN003365, assessed by frequency of adverse events, including worsening of medical conditions/diseases | From Day 1 Cycle 1 through the last day of treatment with ZEN003365 (12 weeks, average)
Dose escalation stage - To characterize the DLTs of orally administered ZEN003365, using NCI CTCAE v4.03 | The first 25 days of at least 12 doses of ZEN003365
Dose expansion stage - Preliminary evidence of the antitumor activity of orally administered ZEN003365 in selected patients, assessed by objective response, duration of objective response and progression-free survival | From Day 1 Cycle 1 through the last day of treatment with ZEN003365 (12 weeks, average)
Dose expansion stage - The safety of orally administered ZEN003365, at the dose chosen based upon the dose escalation stage, assessed by frequency of adverse events, including worsening of medical conditions/diseases | From Day 1 Cycle 1 through the last day of treatment with ZEN003365 (12 weeks, average)

SECONDARY OUTCOMES:
Dose escalation stage - To characterize the pharmacokinetics (PK) of orally administered ZEN003365 in patients, using the following parameters: AUC, Tmax, Cmax, Cmin, pre-dose concentration, and accumulation ratio | From Day 1 Cycle 1 through the last day of treatment with ZEN003365 (12 weeks, average)
Dose expansion stage - To characterize the PK of orally administered ZEN003365, at the dose chosen based upon the dose escalation stage, using the following parameters: AUC, Tmax, Cmax, Cmin, pre-dose concentration, and accumulation ratio | From Screening Visit through 40 days after the last day of treatment with ZEN003365 (19 weeks, average)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee